CLINICAL TRIAL: NCT01689285
Title: Bioequivalence Study in Healthy Volunteers of a New Paediatric Formulation of Valacyclovir Used for Prophylaxis and Treatment of VZV and HSV Infections in Children, Phase I (VALID-I)
Brief Title: Bioequivalence Study in Healthy Volunteers of a New Paediatric Formulation of Valacyclovir
Acronym: VALID-I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF 11.04
Record Dates: First submitted 2012-09-17; First posted 2012-09-21 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Varicella Zoster Virus Infection; Herpes Simplex Virus Infection
Keywords: bioequivalence; pharmacokinetics; valacyclovir; paediatric formulation
MeSH Terms: conditions — Varicella Zoster Virus Infection; Herpes Simplex | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- valacyclovir tablet (Active Comparator): Administration of 500 mg once daily on day 1 (group A) or on day 8 (group B)
  Interventions: Drug: valacyclovir tablet
- valacyclovir oral solution (Experimental): Administration of 500 mg once daily on day 1 (group B) or on day 8 (group A)
  Interventions: Drug: valacyclovir oral solution

INTERVENTIONS:
Drug: valacyclovir tablet — 16 healthy adult volunteers (18-55 yr) will be exposed to one tablet
  Other Names: Zelitrex
  Arms: valacyclovir tablet
Drug: valacyclovir oral solution — 16 healthy adult volunteers (18-55 yr) will be exposed to 10 ml once
  Arms: valacyclovir oral solution

SUMMARY:
A new paediatric formulation (oral liquid) has been developed for flexible and accurate dosing of valacyclovir in children. To establish the bioavailability of this new formulation, healthy volunteers will be exposed to the new formulation and to valacyclovir tablets. The concentration of valacyclovir in their blood after exposure to the oral liquid will be measured and compared to the tablet.

DETAILED DESCRIPTION:
Bioequivalence of the new valcyclovir formulation will be tested according to the EMA guideline for bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 and not older than 55 years of age at screening.
* Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to the first dosing
* Subject has a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2, extremes included.
* Subject has signed the Informed Consent Form prior to screening evaluations.
* Subject is in good age-appropriate health condition as established by medical history, physical examination, electrocardiography, results of biochemistry, haematology and urinalysis testing within 4 weeks prior to the first dose. Results of biochemistry, haematology and urinalysis testing should be within the laboratory's reference ranges (see Appendix A). If laboratory results are not within the reference ranges, the subject is included on condition that the investigator judges that the deviations are not clinically relevant. This should be clearly recorded.
* Subject has a normal blood pressure and pulse rate, according to the investigator's judgement.
* Female subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or is of childbearing potential with adequate contraception (e.g. hysterectomy, bilateral tubal ligation, (nonhormonal) intrauterine device, total abstinence, double barrier methods, vasectomized partner).

Exclusion Criteria:

* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Positive HIV, hepatitis B or C test.
* Therapy with any drug (for two weeks preceding dosing), except for acetaminophen.
* Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), gastro-intestinal disorders, renal and hepatic disorders, hormonal disorders (especially diabetes mellitus), coagulation disorders.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* History of or current abuse of drugs, alcohol or solvents.
* Inability to understand the nature and extent of the trial and the procedures required.
* Participation in a drug trial within 60 days prior to the first dose.
* Donation of blood within 60 days prior to the first dose.
* Febrile illness within 3 days before the first dose.
* Pregnant female (as confirmed by an HCG test performed less than 4 weeks before the first dose) or breast-feeding female.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Ratios and 90% confidence intervals of pharmacokinetic parameters of acyclovir taken as valacyclovir tablet or oral solution | up to 8 days
  bioequivalence will be determined by comparing AUC0-inf, Cmax and tmax of both formulations in healthy adult volunteers.

SECONDARY OUTCOMES:
Determine the safety profile of a single dose of valacyclovir oral solution | day 1 and 8
  healthy volunteers will be interviewed for adverse events, laboratory safety assessments will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Bas Schouwenberg, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Result] Bastiaans DE, Bartels-Wilmer CM, Colbers AP, Heijens CA, Velthoven-Graafland K, Smeets OS, Vink N, Harbers VE, Warris A, Burger DM. A new paediatric formulation of valaciclovir: development and bioequivalence assessment. Arch Dis Child. 2016 Oct;101(10):971-2. doi: 10.1136/archdischild-2015-310266. Epub 2016 May 9. No abstract available. PMID 27162003